CLINICAL TRIAL: NCT03207984
Title: Xenogeneic Collagen Matrix and Connective Tissue Graft Comparison for Multiple Gingival Recessions in Esthetic Areas: A Non-inferiority Clinical Trial
Brief Title: Comparison Between Connective Graft and Xenogeneic Matrix, in Patients With Multiple Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Principal Investigator, Raphaella Coelho Michel, Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9075852
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Gingival Recession, Generalized
Keywords: Gingival Recession; Collagen Matrix; Periodontics
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control SCTG (Active Comparator): Root coverage surgery with subepithelial connective tissue graft to an extensive treat multiple gingival recessions in aesthetic areas
  Interventions: Procedure: Root coverage surgery
- Test CM (Experimental): Root coverage surgery with Mucograft® collagen matrix to treat an extensive multiple gingival recessions in aesthetic areas
  Interventions: Procedure: Root coverage surgery

INTERVENTIONS:
Procedure: Root coverage surgery — Periodontal plastic surgery aiming the treatment of multiple gingival recessions in aesthetics areas with SCTG and CM

SUMMARY:
Subepithelial connective tissue graft (SCTG) is considered the gold standard for root coverage treatment. However, it is associated with postoperative morbidity, limited amount of donor tissue, and longer surgical time. Thus, the search for a tissue substitute for SCTG is increasing. Currently, one of the possible autogenous soft tissue substitutes found in the market is the Mucograft® xenogeneic matrix (CM). The results with the use of MC are very promising, both for root coverage as well as for the gain of keratinized tissue. The present study consists of a parallel randomized clinical trial to compare SCTG (control group) and CM (test group) in the treatment of Miller's class I and II gingival recessions, multiple in aesthetic areas (upper central incisors, Lateral and canine).

DETAILED DESCRIPTION:
Obtaining an aesthetic smile is one of the main reasons for the patient's demand for dental treatment, especially when it comes to gingival recession. However, there is a lack of evidence in the literature explaining the most appropriate type of treatment for multiple recessions in aesthetic areas. For unitary gingival recessions, the subepithelial connective tissue graft (SCTG) is considered the gold standard because it presents greater predictability for root coverage. However, it is associated with postoperative morbidity, limited amount of donor tissue, and longer surgical time. Thus, the search for a tissue substitute for SCTG is increasing. Currently, one of the possible autogenous soft tissue substitutes found in the market is the Mucograft® xenogeneic matrix (CM). The results with the use of CM are very promising, both for root coverage as well as for the gain of keratinized mucosa. The present study will consist of a double-blind parallel randomized clinical trial to compare SCTG (control group) and CM (test group) in the treatment of Miller's class I and II gingival recessions, multiple in aesthetic areas (central incisors, Lateral, upper canine). All measurements will be evaluated initially and in the periods of 3, 6, and 12 months after the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of multiple gingival recessions ≥ 2 mm, only in aesthetic areas (upper central and lateral incisive, and canine);
* Miller class I and II gingival recession areas
* Non-abrasive, erosive, or carious root surfaces
* Unrotated, non-extruded, and non-movable teeth
* Systemically healthy patients without contraindication to periodontal surgical procedures

Exclusion Criteria:

* Smokers
* Pregnant women and infants
* Patients with a history of periodontal disease or recurrent abscess formation
* Patients previously submitted to surgical procedures for root coverage
* Patients taking anti-convulsant drugs
* Antihypertensives, contraceptives or immunosuppressors
* Patients with low oral hygiene (plaque and bleeding index over 20%)

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Gingival recession depth (GRD) | one year
  Distance in millimeters from ECJ to gingival margin at three points (mesial, center and distal); Distance from cemento-enamel junction to gingival margin = 0 mm

SECONDARY OUTCOMES:
Keratinized mucosa width | year
  Keratinized mucosa width measured with a periodontal probe in millimeters Ideal if keratinized mucosa width > 5mm
Dentin hypersensitivity | year
  Dentin hypersensitivity measured by applying an air jet on teeth and patient fills up a visual analogue scale Ideal if scale = 0

OTHER OUTCOMES:
Complete root coverage | year
  Assessed in which the gingival margin was at or above the cementoenamel junction (CEJ)
Probing Depth (PD) | year
  Distance in millimeters from the gingival margin to the bottom of the gingival sulcus at three points (mesial, center and distal)
Clinical attachment level loss (CAL) | year
  Measured in millimeters from the bottom of the periodontal pocket to the cementoenamel junction at three sites per tooth (mesial, center and distal)
Soft tissue thickness (STT) | year
  Determined at 2mm apical the gingival margin at the central buccal site with anesthetic needle and endodontic stop and digital pachymeter

CONTACTS AND LOCATIONS:
Overall Officials: Raphaella C Michel, PhD, Principal Investigator — University of São Paulo, Bauru School of Dentistry
Locations (1):
- Raphaella C Michel, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGuire MK, Scheyer ET. Xenogeneic collagen matrix with coronally advanced flap compared to connective tissue with coronally advanced flap for the treatment of dehiscence-type recession defects. J Periodontol. 2010 Aug;81(8):1108-17. doi: 10.1902/jop.2010.090698. PMID 20350159
- [Background] Cardaropoli D, Tamagnone L, Roffredo A, Gaveglio L. Treatment of gingival recession defects using coronally advanced flap with a porcine collagen matrix compared to coronally advanced flap with connective tissue graft: a randomized controlled clinical trial. J Periodontol. 2012 Mar;83(3):321-8. doi: 10.1902/jop.2011.110215. Epub 2011 Jul 1. PMID 21721988